CLINICAL TRIAL: NCT06968676
Title: Effects of Mixed Reality on Manipulative Skills, Functionality and Quality of Life in People With Multiple Sclerosis. A Randomized Controlled Trial (VIRTUAL-DOMUS)
Brief Title: Mixed Reality for Upper Limb Rehabilitation in People With Multiple Sclerosis (VIRTUALDOMUS)
Acronym: VIRTUALDOMUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Roberto Cano de la Cuerda, PT, PhD. Full Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UniversidadRJC2
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Mixed reality; Upper limb; Rehabilitation; Manipulative skills; Functionality; Quality of life
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Rehabilitation treatment. We do not use drugs or vaccines.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator who will randomize the sample will be external to any intervention. The evaluators will be external to any intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional upper limb training (Active Comparator): Conventional physical therapy exercises for the upper limb, including joint mobilization of the shoulder, elbow, wrist and fingers, forearm and hand muscle strengthening exercises, gross and fine motor work and functional task practice with the aim of mimicking the movements included in the settings specifically designed for experimental intervention
  Interventions: Other: Conventional Upper Limb Treatment
- Mixed reality (Experimental): The experimental group will receive the same conventional physiotherapy treatment plus an extended reality protocol, using Meta Quest 3.0. glasses, by retraining on tasks specifically designed for this project and linked to the specific locations (kitchen, bathroom, living room, bedroom and garden-terrace; see Annexes, page 2, "Recommendations on the development of mixed reality environments"). The intervention will be carried out by a physiotherapist skilled in the use of the technology. The patient's initial position will be seated in front of a table at mid-trunk height, with the elbow at 90° of flexion and the forearm in neutral pronation-supination. The therapist will provide manual assistance as needed, moving to upright sitting or standing positions as the protocol progresses and as tasks require, and work will be done bilaterally.
  Interventions: Other: Experimental intervention with mixed reality

INTERVENTIONS:
Other: Conventional Upper Limb Treatment — Control group (CG) will receive two 60-minute sessions per week for a period of ten weeks (a total of 20 sessions per group). The CG will receive a specific conventional physiotherapy intervention by a physiotherapist with expertise in the care of people with MS. This intervention will be based on conventional physiotherapy exercises [23], including shoulder, elbow, wrist and finger joint mobilization, forearm and hand muscle strengthening exercises, gross and fine motor work and functional task practice with the aim of mimicking the movements included in the settings specifically designed for the experimental intervention.
  Arms: Conventional upper limb training
Other: Experimental intervention with mixed reality — Experimental group will receive the same conventional physiotherapy treatment (40 minutes) in addition to a mixed reality protocol, using Meta Quest 3.0. glasses (20 minutes), by retraining on tasks specifically designed for this project and linked to the specific locations (kitchen, bathroom, living room, bedroom and garden-terrace. The intervention will be carried out by a physiotherapist skilled in the use of the technology. The patient's initial position will be seated facing a table at mid-trunk height, with the elbow at 90° of flexion and the forearm in neutral pronation-supination. The therapist will provide manual assistance as needed, moving to upright-high seated or standing positions as the protocol progresses and as tasks require, and work will be done bilaterally.
  Arms: Mixed reality

SUMMARY:
Although virtual reality has attracted the attention of health professionals and neurorehabilitation field, research about mixed reality (MR) in people with neurological disorders, particularly multiple sclerosis (MS), is very limited. Furthermore, to our knowledge, studies about the effects of MR in upper limb (muscle strength and fatigability, coordination and dexterity, functionality and quality of life) in people with MS are nonexistent.

The main objective of our study are:

To know the clinical effects of mixed reality environments and re-training activities linked to their spaces (kitchen, bathroom, living room, bedroom and terrace-garden), designed for the treatment of upper limb impairments in people with MS, in combination with a conventional physiotherapy program, on manipulative skills, functionality and quality of life in people with MS.

The secundary objectives are:

To study the clinical effects on range of motion, muscle strength, coordination and manual dexterity, fatigue, functionality and quality of life in people with MS.

To analyze satisfaction and adherence to treatment, the occurrence of adverse effects and the level of workload perceived by participants.

A double-blind randomized controlled trial is proposed. The sample will be randomly divided into two groups: the experimental group will receive treatment based on mixed reality for MMSS, designed by the research team and using Meta Quest 3.0 glasses, in combination with conventional physiotherapy; and the control group will receive the same conventional therapy. Both groups will receive 2 sessions/week, 60min/session, for 10 weeks. The mixed reality environments to be designed will be a kitchen, a bathroom, a living room, a bedroom and a terrace-garden, with the tasks to be performed in each location. The pre, post-treatment and one-month follow-up outcome measures will be: range of motion, manual grip strength, manual dexterity, fatigue, functionality, quality of life, satisfaction with the technology, adherence, adverse effects and perceived workload. A statistical comparison study will be carried out establishing as an inter-subject factor the group parameter and as intra-subject factors each of the measurements and the treated side.

DETAILED DESCRIPTION:
MS is a neurological pathology that currently affects approximately 36 people per 100,000 inhabitants (2.8 million people affected in the world) and has various clinical manifestations, such as alterations in balance and coordination, fatigue or alterations in sensitivity, with alterations in the motor control of the MMSS being one of the main problems faced by people with MS from the time of diagnosis, the main consequence of which is an alteration in their ability to perform ADLs, reducing their quality of life.

Although new drugs aimed at modifying the course of the disease have appeared in recent years, there is currently no curative treatment for MS. For this reason, pharmacological therapy is complemented by rehabilitative treatment in order to maintain functional capacity and favor adaptation to the changes produced by the evolution of the disease itself. However, conventional rehabilitation treatment of people with MS is sometimes referred to as systematic, so that patients may lose motivation and adherence to it. This is why in recent years new intervention strategies have been introduced, such as VR, which encourage patient motivation through the practice of functional tasks in virtual environments that provide feedback on the results obtained and the possibility of increasing repetitions and work intensity through simulated ADL training.

The development of these technologies has offered professionals working in the field of neurological rehabilitation to extend the care of MS patients as a complement to their conventional rehabilitation program, reaching a higher intensity of treatment and sometimes at a sustainable cost. However, studies on the effects of VR on manipulative skills in people with MS are still scarce and, to our knowledge, quality studies proposing the use of mixed reality as a tool for the treatment of MMSS impairments in people with MS are nonexistent.

For the reasons described above, an RCT is justified to investigate the effects of the application of a treatment protocol through mixed reality environments that simulate the re-training of activities in the locations of a house (from the Latin, "domus") and, therefore, facilitate its transfer from learning to the real world, on manipulative skills, functionality and quality of life in people with MS (VIRTUAL-DOMUS), following international recommendations on the design of virtual environments for therapeutic purposes in neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

->18 years of age.

* Diagnosis of MS according to McDonald criteria (53) with a time of evolution longer than two years.
* Assessment on the Kurtzke Multiple Sclerosis Disability Status Scale (EDSS) with a score between 2. 0 (minimal disability in one section of the FS (at least one with a score of 2).) to 7.0 (unable to walk more than a few steps, even with assistance, basically confined to wheelchair and able to transfer from wheelchair to another place, or can manage to go to the toilet for 12 hours a day) .
* Stable medical treatment for at least six months prior to surgery.
* Upper extremity muscle tone no greater than 2 points (moderate hypertonia, increased muscle tone during most of the arc of motion, but can passively move the affected part with ease) on the modified Ashworth Scale.
* Muscle balance equal to or greater than 3 in the upper extremity.
* Score less than or equal to 4 points on the "Pyramidal Function" section of the EDSS functional scale.
* Absence of cognitive impairment, with ability to understand instructions and score equal to or greater than 24 on the Minimental Test.

A- score equal to or less than 2 points on the "Mental Functions" section of the EDSS.

Exclusion Criteria:

* Diagnosis of a neurological disease or musculoskeletal disorder other than MS.
* Diagnosis of a cardiovascular, respiratory or metabolic disease or other conditions that may interfere with this study.
* Having suffered an exacerbation or hospitalization in the last 3 months before starting the assessment protocol, or during the therapeutic intervention process.
* Having received a course of steroids, intravenous or oral, 6 months prior to the start of the assessment protocol and within the intervention period of the study duration.
* Having received treatment with botulinum toxin in the 6 months prior to the start of the study.
* A score higher than 2 points on the modified Ashworth scale.
* Cognitive or language impairment that prevents adequate communication or comprehension.
* The presence of visual disturbances not corrected by ocular devices; or a history of photosensitive epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Isometric prehensile hand strength (Kg) | Up to 10 weeks
  Isometric prehensile hand strength: measured by the JAMAR® fist dynamometer. The JAMAR® dynamometer has been widely cited and is considered the gold standard for the assessment of fist strength. Three measurements of the maximum voluntary maximum isometric contraction (MVC) will be taken with each hand, always starting with the least affected hand; once the three measurements have been taken, the mean of these will be obtained.
  Major values (Kg) means a higher hand grip strengh (there is not a maximum).

SECONDARY OUTCOMES:
Isometric pincer force (Kg) | Up to 10 weeks
  Isometric pincer force: a Baseline Pinch Gauge® will be used to assess 3 different types of pinch: terminal opposition grip, in which the anterior and distal face of the first finger contacts the anterior face of the dynamometer, anterior and distal face of the second finger contacts the posterior face of the dynamometer; pulpolateral grip, in which the anterior face of the distal phalanx of the first finger contacts the anterior face of the dynamometer, radial edge of the second finger contacts the posterior face of the dynamometer; tridigital press of the first three fingers, in which the anterior and distal face of the first finger contacts the posterior face of the dynamometer, anterior and distal face of the second and third finger contacts the anterior face of the dynamometer. As in the previous test, 3 measurements will be taken and the average score will be obtained.
  Major values (Kg) means a better pincer force strengh (there is not a maximum)
Gross coordination for the upper limb (Block and Box; number of cubes) | Up to 10 weeks
  Box and Block Test (BBT): it will be used to assess coordination and manual dexterity. The patient is seated with the tool, a wooden box divided into two identical halves inside which there are 150 wooden cubes of 2.5 cm of different colors, in front of his midline. The patient has to move as many cubes as possible from one half of the box to the other in 60 seconds. The test is performed first with the dominant hand and then with the non-dominant hand. It is a standardized tool for the measurement of the gross function of the MMSS, having been validated by gender and age in healthy subjects, in turn, it shows a low ceiling and floor effect in people with MS.
  pincer force A higher number of cubes (there is not a maximun) indicate a better coordination of the upper limb.
Fine coordination for the upper limb (NHPT; time in seconds) | Up to 10 weeks
  Nine Hole Peg Test (NHPT): this test will be used to assess the function of the MMSS, in particular the fine motor skills of the hand. The tool will be placed in front of the subject's midline, the subject will have to insert the 9 pegs, one at a time, into the 9 holes of a board and then remove them, again one at a time, in the shortest possible time; first with the dominant hand, and then the non-dominant hand, the hand that is not being assessed can hold the board to provide stability. The score is the time in seconds required to insert and remove all the pins. It shows excellent test-retest, inter-rater and inter-rater reliability and adequate internal consistency.
  Lower time in seconds (s) (not specificated the minimum) in the test indicates a better fine coordination.
Functional status of the upper limb (ABILHAND) | Up to 10 weeks
  Abilhand: is a self-administered questionnaire to assess the person's manual dexterity, defining this as the ability to perform a series of tasks, regardless of the strategies applied to achieve it. The questionnaire contains 23 items scored from 0 to 2, which correspond to various ADL tasks; the patient will mark the degree of difficulty he or she refers to when performing the activities. The score can range from 0 to 46 points, the higher the score, the better the manual dexterity. Its inter- and intra-rater reliability, internal consistency and construct validity are excellent.
  A higher score (maximun 46 points) indicates a better functionality.
Quality of life (MSIS-29) | Up to 10 weeks
  Multiple Sclerosis Impact Scale (MSIS-29): is a self-applied scale on the impact of the disease on the patient's life in the two weeks prior to performing. It presents 29 questions of which 20 assess the physical aspects of MS and 9 assess the psychosocial aspects. The physical sphere has been proven to have high internal consistency and good construct validity, while the cognitive sphere has good internal consistency.
  A higher score (maximun 29 points) indicates a better quality of life.
Satisfaction (CSQ8) | Up to 10 weeks
  CSQ8: self-completed questionnaire with eight dimensions measuring satisfaction with the care and treatment received. The total score is 32 points, where maximum scores indicate higher satisfaction. Dimensions related to satisfaction with the training modality and tool used (entertainment, ease of use, accessibility, among others), the professional who applies it (clear explanation, availability, adaptability, among others) or recommendation to other patients will be evaluated.A higher score (maximun 32 points) indicates a better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cano de la Cuerda, PhD, Principal Investigator — Universidad Rey Juan Carlos

IPD SHARING:
Plan to Share IPD: No